CLINICAL TRIAL: NCT01768143
Title: A Reliable and Valid Assessment of Nurse Administered Propofol Sedation (NAPS) Performance.
Brief Title: Assessment of NAPS Performance.
Acronym: NAPSAT
Status: Completed | Type: Observational
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Sponsor
Other Study IDs: SPAT-003
Record Dates: First submitted 2013-01-09; First posted 2013-01-15 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2013-09

CONDITIONS: Competence in Propofol Sedation for Endoscopy
Keywords: Propofol; Sedation; Endoscopy; nonanesthesiologist

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Nurse Trainees: unexperienced endoscopy nurses
  Interventions: Behavioral: unexperienced endoscopy nurses
- Nurse Experts: Educated endoscopy Nurses
  Interventions: Behavioral: Experienced endoscopy nurses

INTERVENTIONS:
Behavioral: unexperienced endoscopy nurses
  Groups: Nurse Trainees
Behavioral: Experienced endoscopy nurses
  Groups: Nurse Experts

SUMMARY:
To measure competencies in propofol sedation for endoscopic procedures (NAPS)through development, test and validation of a reliable assessment tool in a simulator setting.

Hypothesis: That the tool will demonstrate content and construct validity, ie. enable reliable measuring of necessary competencies of different levels in a reproducible way.

ELIGIBILITY:
Inclusion Criteria:

* eligible nurses, written informed consent.

Exclusion Criteria:

* Prior anesthesia or ICU experience

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Endoscopy nurses of different competencylevel
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2013-01; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Assessed sedation performance score | 6 months
  A Total of 12 Global Rating Scores and 2 checklist scores on hands on performance in a simulation setting and a theoretical Multiple Choice questionnaire. The performance score is decided by independent raters who review performances on video.

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev Hospital, Gastroenheden, Copenhagen, Herlev, Herlev, Denmark